CLINICAL TRIAL: NCT05361057
Title: A Prospective, Single Arm, Multicenter Clinical Study to Evaluate the Efficacy of Venetoclax Combined With Azacytidine or DA Regimen in Prevention the Relapse of Consecutive MRD Positive AML Patients
Brief Title: Efficacy of Venetoclax Based Regimen in Prevention Relapse of Consecutive MRD Positive AML Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The research center has conducted a more comprehensive study.
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022006
Record Dates: First submitted 2022-03-14; First posted 2022-05-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia; Measurable Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- venetoclax pluse azacitidine arm (Experimental): azacytidine 75 mg/m2 d1-7，venetoclax: 100mg d1, 200mg d2, 400mg d3-21
  Interventions: Drug: Venetoclax, Azacitidine
- venetoclax pluse DA arm (Active Comparator): daunorubicin：45mg/m2 d1-2, cytarabine:100mg/ m2 d1-5, venetoclax: 100mg d1, 200mg d2, 400mg d3-14
  Interventions: Drug: Venetoclax, daunorubicin, cytarabine

INTERVENTIONS:
Drug: Venetoclax, Azacitidine — The patients were administrated with azacytidine 75 mg/m2 d1-7，venetoclax: 100mg d1, 200mg d2, 400mg d3-21;
  Arms: venetoclax pluse azacitidine arm
Drug: Venetoclax, daunorubicin, cytarabine — The patients were administrated with daunorubicin：45mg/m2 d1-2, cytarabine:100mg/ m2 d1-5, venetoclax: 100mg d1, 200mg d2, 400mg d3-14
  Arms: venetoclax pluse DA arm

SUMMARY:
Measurable disease (MRD) plays an important role in the therapeutic efficacy and prognosis of acute myeloid leukemia (AML). Studies show that persistent MRD positivity after induction indicates that the patient has a higher risk of recurrence. Even if the patient is assessed as a low risk group, once there is persistent MRD positive, Allogeneic hematopoietic stem cell transplantation (allo HSCT) or clinical trials should be considered to improve the overall survival of patients. However, some patients cannot accept allo HSCT due to economic reasons or lack of suitable donors. How to prolong the recurrence free survival of these patients is still a great challenge. Platzbecker et al. applied azacytidine (AZA) monotherapy to AML patients with continuous MRD positive after combined chemotherapy. The results showed that the preemptive treatment of AZA could prevent or significantly delay the hematological relapse of MDS or AML patients with MRD positive. In addition, the application of venetoclax has significantly changed the therapeutic prospect of AML and provided new opportunities. Studies have shown that venetoclax can enhance the activity of anti HMA, cytarabine, idarubicin and other drugs. The curative effect of venetoclax combined with AZA in the treatment of elderly AML patients who are not suitable for intensive treatment is better than that of single AZA regimen, and the negative rate of MRD after induction treatment of venetoclax combined with HMA is higher (54-81%). Therefore, the investigators believe that for patients who continue to be MRD positive after induction and consolidation treatment, venetoclax based regimen may be an effective preemptive treatment regimen, which can prolong the relapse free time and overall survival of these patients

DETAILED DESCRIPTION:
In the study, 40 patients will be enrolled and treated with venotoclax combined AZA and DA regimen. Patients receive major response will be given venotoclax combined AZA regimen as maintenance treatment. The primary endpoint was 6 month relapse-free survival. Measurable residual disease (MRD) will be detected at the beginning of the therapy and after the therapy. The adverse effect will also be explored.

Preemptive chemotherapy: regimen 1: azacytidine 75 mg/m2 d1-7，venetoclax: 100mg d1, 200mg d2, 400mg d3-21; regimen 2: daunorubicin：45mg/m2 d1-2, cytarabine:100mg/ m2 d1-5, venetoclax: 100mg d1, 200mg d2, 400mg d3-14; maintenance therapy: patient in regimen 1 group: azacytidine 75 mg/m2 d1-7，venetoclax: 400mg d1-14, for 4 cycles, patients in regimen 2 group: azacytidine 75 mg/m2 d1-7，venetoclax: 400mg d1-14, for 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed acute myeloid leukemia
2. Received chemotherapy within 24 months and has completed the consolidation treatment plan
3. In complete remission
4. With MRD positive: abnormal myeloid cells in bone marrow ≥ 0.1%, or NPM1 gene mutation and other fusion gene positive(RUNX 1-RUNX1T 1、CBFB-MYH11 and DEK-NUP214), the PCR quantification ≥1%.
5. Age≥ 18 years #male or female
6. ECOG-PS score 0-2
7. Aboratory tests#within 7 days before chemotherapy# 1). Serum total bilirubin≤1.5xULN# 2). Serum AST and ALT≤2.5xULN 3). Serum creatinine≤2xULN# 4). Cardiac enzymes≤2xULN 5). Ejection fraction >50% by ECHO#
8. Written informed consent

Exclusion Criteria:

1. Hematological relapse (the proportion of blast cells in bone marrow is greater than 5%)
2. Receive hematopoietic stem cell transplantation within 4 weeks
3. APL
4. Have been treated with venetoclax in the past 6 months (who can be enrolled after stopping for more than 6 months)
5. Suffering from malignant tumors of other organs (those requiring treatment)
6. Pregnant or lactating women
7. Active heart diseases
8. Severe active infection
9. Unfit for enrollment evaluated by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
relapse free survival | 6 months
  survival from the preemptive therapy to relapse

SECONDARY OUTCOMES:
major response | 3 months
  The MRD level turns negative or the specific value decreases by 1 order of magnitude
overall survival | 1 year
  duration from enrollment to death or loss of followup
relapse free survival | 12 months
  survival from the preemptive therapy to relapse

CONTACTS AND LOCATIONS:
Locations (1):
- HBDH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No